CLINICAL TRIAL: NCT01732224
Title: A Prospective Randomized Controlled Study to Compare the Efficacy of Combined Tenofovir Plus Telbuvidine vs Tenofovir Alone in Patients With Spontaneous Reactivation of Hepatitis B.
Brief Title: To Compare the Efficacy of Combined Tenofovir Plus Telbivudine vs Tenofovir Alone in Patients With Spontaneous Reactivation of Hepatitis B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-HBV Reactivation-01
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2012-11

CONDITIONS: Spontaneous Reactivation of Hepatitis B
MeSH Terms: interventions — Tenofovir; Telbivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tenofovir + Telbivudine (Experimental): Tenofovir (300 mg/day) plus telbivudine (600 mg/day).
  Interventions: Drug: Tenofovir
- Tenofovir (Active Comparator): In tenofovir arm subjects will receive tenofovir (300 mg) once daily.
  Interventions: Drug: Tenofovir + Telbivudine

INTERVENTIONS:
Drug: Tenofovir + Telbivudine — Tenofovir (300 mg/day) plus telbivudine (600 mg/day).
  Arms: Tenofovir
Drug: Tenofovir — In tenofovir arm subjects will receive tenofovir (300 mg) once daily.
  Arms: Tenofovir + Telbivudine

SUMMARY:
The relevant data will be prospectively collected included patient demographics, clinical, all laboratory variables including virological tests, genotyping by direct sequencing, abdominal ultrasound, and upper gastrointestinal (GI) endoscopy. Trans jugular liver biopsy (TJLB) and hepatic venous pressure gradient (HVPG) will be done in patients when it was not evident whether the underlying liver disease was chronic based on clinical, biochemical, radiological investigations, and upper GI endoscopy. Severity of the liver disease will be assessed by Child-Turcotte Pugh score (CTP) and model for end stage liver disease (MELD) score.

ELIGIBILITY:
Inclusion Criteria:

* Reactivation of CHB characterized by a rise in ALT level >5 times upper limit of normal along with HBV DNA level >10^5 copies/ mL (> 1.8 X 10^4 IU/mL).

Exclusion Criteria:

1. Superinfection with other viruses (hepatitis E, A, D, or C)
2. other causes of chronic liver failure
3. coexistent hepatocellular carcinoma (HCC)
4. portal vein thrombosis
5. coexistent renal impairment
6. pregnancy
7. coinfection with human immunodeficiency virus (HIV)
8. patients who had received a previous course of any antiviral, immunomodulator or cytotoxic/immunosuppressive therapy for chronic hepatitis or other illness within at least the preceding 12 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2012-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Survival | 1 and 3 months

SECONDARY OUTCOMES:
Reduction in HBV DNA. | 7 days, 15 days, 1 month and 3 month
Drug(s) related adverse effects/ side effects | 1 and 3 months
Improvement in CTP and MELD scores | 1 and 3 months
Alteration of renal functions | 1 and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Shiv Kumar Sarin, DM, Principal Investigator — Institute of Liver & Biliary Sciences (ILBS).
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India